CLINICAL TRIAL: NCT01233375
Title: A Phase II, Open-Label, Multicenter Study to Evaluate the Antitumor Efficacy of CO-1.01 for Infusion as Second-Line Therapy for Gemcitabine- Refractory Patients With Stage IV Pancreatic Adenocarcinoma and No Tumor hENT1 Expression
Brief Title: Study to Evaluate Efficacy of CO-1.01 as Second Line Therapy for Gemcitabine-Refractory Stage IV Pancreatic Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-101-003
Record Dates: First submitted 2010-10-26; First posted 2010-11-03 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: cancer; metastatic; pancreatic; pancreas; adenocarcinoma; gemcitabine; human equilibrative nucleoside transporter-1 (hENT1); CO-1.01; CO-101; CO101; Stage 4; Stage IV; Gemcitabine-Refractory; Second-Line Therapy
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CO-1.01 (Experimental)
  Interventions: Drug: CO-1.01

INTERVENTIONS:
Drug: CO-1.01 — 1250 mg/m2/day administered on Days 1, 8, and 15 in 4-week treatment cycles.
  Patients who have SD or better at the Week 8 assessment and who adequately tolerated the first 2 cycles of treatment may continue CO-1.01 at the same or an increased dose (1400 mg/m2) for Cycle 3 and subsequent cycles.

SUMMARY:
The purpose of this study is to determine whether CO-1.01 is safe and effective for treating metastatic pancreatic cancer that did not respond to gemcitabine.

DETAILED DESCRIPTION:
Pancreatic tumors with low hENT1 expression may show less benefit from gemcitabine compared with those with higher expression of this nucleoside transporter. Nonclinical studies indicate that CO-1.01, a gemcitabine derivative, is effective independent of such transporters. Thus patients with low or no meaningful expression of hENT1 who failed to respond to gemcitabine might derive benefit from CO1.01 before needing alternative (combination) chemotherapy. Furthermore, the PK profiles of CO-1.01 and gemcitabine are dissimilar and this may confer additional clinical benefit on CO1.01.

ELIGIBILITY:
Inclusion Criteria:

1. Gemcitabine-refractory metastatic ductal adenocarcinoma of the pancreas

   * At least 1 measurable lesion according to RECIST 1.1 criteria
   * Computerized tomography (CT) scan ≤ 28 days prior to CO-1.01
   * First-line treatment included at least 3 doses of gemcitabine (as monotherapy or combination therapy) with the last dose administered at least 2 weeks prior to CO 1.01
   * Radiological best response of disease progression after 1st-line treatment (no radiological stable disease or better allowed at any time)
   * Patients who experienced progressive disease during (neo)-adjuvant gemcitabine-based therapy are also eligible
   * Patients who have completed previous adjuvant therapy without progression, then subsequently have a radiological best response of disease progression on 1st line gemcitabine for metastatic disease are eligible
2. No hENT1 expression in primary or metastatic tumor sample, confirmed with IHC by a core pathology laboratory prior to study entry also eligible
3. Performance Status (ECOG) 0 or 1
4. Age ≥18 years
5. Palliative radiotherapy (if administered) ≥2 weeks prior to CO-1.01
6. Adequate hematological and biological function, with no residual gemcitabine-related toxicity
7. Written consent on an Institutional Review Board (IRB)-approved IC Form prior to any study-specific evaluation

Exclusion Criteria:

1. Patients who have had stable disease, partial response or complete response to first line gemcitabine-based therapy
2. First-line chemotherapy regimen that does not contain gemcitabine
3. First-line treatment discontinued due to intolerable gemcitabine-induced toxicity
4. Second or subsequent line therapy for advanced disease. Prior exposure to CO-1.01 or prior randomization in a protocol studying CO-1.01 (e.g.,Protocol CO-101-001)
5. Tumor that cannot be evaluated for hENT1 expression or that has hENT1 staining in >50% of cells
6. Symptomatic brain metastases
7. Concomitant treatment with prohibited medications (e.g., concurrent anticancer therapy including other chemotherapy, radiation, hormonal treatment [except corticosteroids and megestrol acetate], or immunotherapy) ≤14 days prior to CO-1.01
8. Exploratory laparotomy, palliative (e.g., bypass) surgery, or other procedures are not allowed <14 days prior to CO-1.01 administration; stenting procedures are permissible at any time prior to dosing; in all cases, the patient must be sufficiently recovered and stable
9. History of allergy to gemcitabine or eggs
10. Females who are pregnant or breastfeeding
11. Refusal to use adequate contraception for fertile patients (females and males during the study and for 6 months after the last dose of CO-1.01)
12. Presence of any serious or unstable concomitant systemic disorder incompatible with the clinical study (e.g., substance abuse, psychiatric disturbance, uncontrolled intercurrent illness including active infection, arterial thrombosis, or symptomatic pulmonary embolism)
13. Any other reason for which the investigator considers the patient should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Disease Control Rate (CR, PR, or SD) using RECIST 1.1 | Every 8 weeks until disease progression

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Every 8 weeks
CA 19-9 response rate | Every 4 weeks
Progression-free survival (PFS) | Every 8 weeks
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Every week
Overall survival (OS) | 3, 6, 9, and 12 months
Median progression-free survival | 3, 6, 9, and 12 months
Median overall survival | 3, 6, 9, and 12 months
Duration of response | Every 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eileen O'Reilly, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (13):
- United States (13):
  - Arizona Cancer Center at University of Arizona, Tucson, Arizona
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Palm Beach Institute / Collaborative Research Group, Boynton Beach, Florida
  - University of Miami, Miami, Florida
  - Piedmont Healthcare Research Institute (PHRI), Atlanta, Georgia
  - Norton Cancer Institute Research Program, Louisville, Kentucky
  - Johns Hopkins Oncology Center, Baltimore, Maryland
  - Massachusetts General Hospital (MGH), Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Columbia University Medical Center, Milstein Hospital, New York, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin